CLINICAL TRIAL: NCT04432909
Title: A Prospective, Multi-centre, Single-blinded Study of UroCAD for Urothelial Carcinoma Diagnosis and Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: RenJi Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Zhejiang Provincial People's Hospital (Other); Tongji Hospital (Other); Tianjin Medical University Second Hospital (Other); Qilu Hospital of Shandong University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Xibei Hospital (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Shuxiong Zeng, Principal Investigator, Changhai Hospital
Other Study IDs: CH-urothelial-cancer-marker
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Urothelial Carcinoma
Keywords: diagnosis; follow-up
MeSH Terms: conditions — Carcinoma, Transitional Cell; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from Urine Exfoliated Cells will be analyzed
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urothelial carcinoma group: Pre-surgery patients with urothelial carcinoma will be the experimental group to determine the sensitivity and specificity of UroCAD analysis, the result will be compared with cytology and FISH test.
  Interventions: Diagnostic Test: The level of CNV
- Non-cancer participants: Patients being treated for other diseases but without any tumor will provide a negative control to provide data for determining the sensitivity and specificity of UroCAD analysis.
  Interventions: Diagnostic Test: The level of CNV

INTERVENTIONS:
Diagnostic Test: The level of CNV — The extracted DNA from morning urine will be analyzed by UroCAD to determine the level of CNV. And the patient will be followed for up to 2 years.
  Other Names: UroCAD test of the urine exfoliated cells

SUMMARY:
Urothelial carcinoma (UC) is common malignancy and is considered to be one of the costliest cancers. The traditional diagnostic methods of UC present with some shortcomings. For example, the specificity of CTU remains low while cystoscopy is invasive and expensive. Therefore, a noninvasive diagnostic method with high accuracy is urgently needed. Our previous study has proved that UroCAD, which is able to detect chromosomal aberrations of the urine exfoliated cells, is a reliable method in diagnosing UC with sensitivity and specificity of 82.5% and 96.9%, respectively. But its potential in UC patient follow-up hasn't been assessed yet and the the accuracy of UroCAD in detecting UC still need to be further validated. The investigators here intended to investigate whether UroCAD can be used in UC patient follow-up and further validate the accuracy of UroCAD in diagnosing UC.

DETAILED DESCRIPTION:
The traditional diagnostic methods of UC include CT urography (CTU) and cystoscopy. To access the upper urinary tract, CTU is commonly used. The sensitivity for detecting upper tract urothelial cancer with CTU has been reported to reach 89%. However, the specificity of CTU is 51% and it cannot get a biopsy sample. Other shortcomings include exposing the patient to high dose of radiation and the contrast material usage may impair the renal function. In the context of diagnosing lower urinary tract cancer, cystoscopy is the "gold standard" diagnostic procedure, which has a sensitivity of 68-83%. But it is invasive, uncomfortable and may miss flat lesions. Furthermore, due to the high recurrence rate of bladder cancer, surveillance of the disease with frequent cystoscopy make it one of the costliest cancers. Therefore, a noninvasive diagnostic method with high accuracy is urgently needed.

Copy number variations (CNVs) refers to the ongoing acquisition of genomic alterations ranging from point mutations to gross chromosomal rearrangements, is a hallmark of cancer which is found in 60-80% of human cancer, and it positively correlates with high tumor stage, poor prognosis, metastasis and therapeutic resistance. Several researches have investigated the value of detecting chromosomal instability with sWGS in either cell-free (cf)DNA or genomic DNA as a noninvasive diagnostic method for cancers and yielded quite fine results. Our previous research has also proved the UroCAD model reached performance of AUC=0.928, with sensitivity, specificity and accuracy of 82.5%, 96.9% and 89.0%, respectively. This test also showed superiority in diagnosing upper tract urothelial cancer compared with urinary cytology test.

Here the investigators intended to conduct a prospective, multicenter, single-blinded research to further validate the value of UroCAD in diagnosing UC and investigate the potential of UroCAD in UC patient follow-up by analyzing the CNV level of patient DNA extracted from urine exfoliated cells and follow UC patient for up to 2 years to determine if there is a correlation between CNV level and patient prognosis. Patient information, which is acquired every 3 months after surgery, including survival status, CNV level in urine exfoliated cells, treatment during this period, medical examination during this period, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with urothelial carcinoma and planned to undergo surgery
* Cancer patient with urine cytology test result
* Cancer patient willing to provide urine sample before the surgery, 3 months after surgery, 6 months after surgery, 12 month after surgery, 15 months after surgery, 18 months after surgery, 21 months after surgery, 24 months after surgery, and willing to provide patient information.
* Participants without any tumor disease and willing to attend the study by providing morning urine.
* Male or female patients aged >= 18 years.
* Participants signed informed consent form.

Exclusion Criteria:

* Age under 18 years
* Individuals unwilling to sign the consent form or unwilling to provide morning urine for test or unwilling to provide the medical record.
* Patient already received suprapubic cystostomy or urethral catheterization.
* Patient with late-stage uremia and need regular dialysis.
* Patient with cancer other than urothelial carcinoma.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with urothelial carcinoma or participants in control group from January 2020 to June 2022 in 10 hospitals including Changhai hospital, Renji hospital, The First Affiliated Hospital of Suchow university, Zhejiang Provincial people's hospital, Tongji hospital, The second hospital of Tianjin medical university, Qilu hospital, Second Affiliated Hospital of Sun Yat-Sen University, Xibei hospital, West China hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of urinalysis by UroCAD analysis | through study completion, an average of 30 months
  number of patients "declared positive" with the UroCAD test among the patients suffered from urothelial carcinoma and number of patients "declared negative" with the UCAD test among the patients without cancer.
Assess the value of UroCAD for urothelial cancer patient follow-up | through study completion, an average of 30 months
  Compare the CNV level with the patient information gathered by follow-up to determine whether there is a correlation between CNV level and patient prognosis or disease progression

SECONDARY OUTCOMES:
Identification of the correlation between the level of CNV and the grade of the tumor sample | through study completion, an average of 30 months
  level of CNV in the urine sample compared with the grade of the tumor confirmed by histopathologic examination
Identification of the correlation between the level of CNV and the stage of the tumor sample | through study completion, an average of 30 months
  level of CNV in the urine sample compared with the stage of the tumor confirmed by histopathologic examination
Comparison of the sensitivity and specificity of the UroCAD analysis versus urine cytology | through study completion, an average of 30 months
  number of patients "declared positive" with the UroCAD analysis versus patients "declared positive" with the urine cytology and number of patients "declared negative" with the UroCAD analysis versus patients " declared negative " with the urine cytology

CONTACTS AND LOCATIONS:
Overall Officials: Chuanliang Xu, M.D.,Ph.D., Study Chair — Changhai Hospital, Shanghai
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will try to protect the information of the included participants

REFERENCES:
- [Background] Wadhwa N, Mathew BB, Jatawa SK, Tiwari A. Genetic instability in urinary bladder cancer: An evolving hallmark. J Postgrad Med. 2013 Oct-Dec;59(4):284-8. doi: 10.4103/0022-3859.123156. PMID 24346386
- [Background] Bakhoum SF, Ngo B, Laughney AM, Cavallo JA, Murphy CJ, Ly P, Shah P, Sriram RK, Watkins TBK, Taunk NK, Duran M, Pauli C, Shaw C, Chadalavada K, Rajasekhar VK, Genovese G, Venkatesan S, Birkbak NJ, McGranahan N, Lundquist M, LaPlant Q, Healey JH, Elemento O, Chung CH, Lee NY, Imielenski M, Nanjangud G, Pe'er D, Cleveland DW, Powell SN, Lammerding J, Swanton C, Cantley LC. Chromosomal instability drives metastasis through a cytosolic DNA response. Nature. 2018 Jan 25;553(7689):467-472. doi: 10.1038/nature25432. Epub 2018 Jan 17. PMID 29342134
- [Background] Liu H, He W, Wang B, Xu K, Han J, Zheng J, Ren J, Shao L, Bo S, Lu S, Lin T, Huang J. MALBAC-based chromosomal imbalance analysis: a novel technique enabling effective non-invasive diagnosis and monitoring of bladder cancer. BMC Cancer. 2018 Jun 15;18(1):659. doi: 10.1186/s12885-018-4571-7. PMID 29907142
- [Background] Hieronymus H, Murali R, Tin A, Yadav K, Abida W, Moller H, Berney D, Scher H, Carver B, Scardino P, Schultz N, Taylor B, Vickers A, Cuzick J, Sawyers CL. Tumor copy number alteration burden is a pan-cancer prognostic factor associated with recurrence and death. Elife. 2018 Sep 4;7:e37294. doi: 10.7554/eLife.37294. PMID 30178746